CLINICAL TRIAL: NCT05318755
Title: China Gender-affirming Hormone Therapy Study in Transgender Men and Women
Brief Title: China Gender-affirming Hormone Therapy Study
Acronym: CGAHT
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Hong Tianpei, Professor, Peking University Third Hospital
Other Study IDs: CGAHT
Record Dates: First submitted 2022-02-16; First posted 2022-04-08 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Transgender; Gender Incongruence
Keywords: Transgender Persons; Gender-affirming Hormone Therapy
MeSH Terms: conditions — Gender Dysphoria | interventions — Testosterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and stool sample will be taken before and during the course of GAHT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- transgender men: People whose sex assigned at birth is female but whose self-identified gender is male.
  Interventions: Drug: GAHT for transgender men
- transgender women: People whose sex assigned at birth is male but whose self-identified gender is female.
  Interventions: Drug: GAHT for transgender women
- Healthy cisgender people: People whose sex assigned at birth corresponds with their self-identified gender.

INTERVENTIONS:
Drug: GAHT for transgender men — Testosterone undecanoate
  Other Names: Testosterone
  Groups: transgender men
Drug: GAHT for transgender women — Estradiol and antiandrogens (Spironolactone or Cyproterone acetate)
  Other Names: Feminizing drugs
  Groups: transgender women

SUMMARY:
Data about transgender medical care, especially the gender-affirming hormone therapy (GAHT) is extremely insufficient in China. Few evidence exists in the physical and psychological effects of the hormonal treatment in Chinese transgender population. CGAHT is designed to describe the social and mental condition of transgender people who are seeking for formal GAHT, and to investigate the physical and psychological effects of GAHT on this population in China.

DETAILED DESCRIPTION:
CGAHT will be conducted in one of the main transgender medical centers in Chinese mainland. Participants who are seeking for the start of GAHT will be enrolled from clinical visitors. Before GAHT, participants will be interviewed with questionaries about their life experience, gender identity and social economic conditions. Evaluations on mental and physical health will be performed at baseline and during the GAHT. Participants will be followed up to 12 months. GAHT will be given to transgender people according to the protocol recommended by the international guideline (doi: 10.1210/jc.2017-01658) .

ELIGIBILITY:
Inclusion Criteria:

* Transgender men and women
* Meet criteria of Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) for gender dysphoria
* Aged between 18 to 40 years
* People desire to start the GAHT
* No previous history of gender-affirming interventions
* Having full ability to make informed consent
* Dextromanual

Exclusion Criteria:

* Disorders of sex development
* Who has fertility demand but have not made fertility preservation
* With contradictions of GAHT
* Comorbid diseases are not under control
* Alcohol or drug abuse
* Hormonal and chromosomal disorders
* History of gender affirming surgery
* Current psychiatric disorders
* History of brain trauma or neurological pathologies
* Current use of medications with psychotropic effects within two weeks (antipsychotic or antiepileptic agents, lithium, benzodiazepines or opioid analgesics)
* Claustrophobia
* Implanted metal and medical devices (pacemakers, ceramic teeth, etc.),
* Tattoos or eyebrow tattooing (heavy metal dye)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men and women are based on self-representation of gender identity
Study Population: 100 transgender men, 100 trangender women, 20 healthy cisgender men and 20 healthy cisgender women
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-04-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Insulin Sensitivity at 12 months | 12 months
  Insulin sensitivity will be assessed with composite insulin sensitivity index (ISI), which is calculated as 10 000/√[(fasting glucose [mg/dL]) ×(fasting insulin [μU/mL]) × (mean glucose [mg/dL]) × (mean insulin [μU/mL])], using 0 min, 60 min, and 120 min values of oral glucose tolerance test (OGTT). Composite ISI will be evaluated at baseline and every 6 months until 12 months of GAHT.
Change from Baseline Beta-cell Function at 12 months | 12 months
  Beta-cell function will be assessed with oral glucose tolerance test-derived disposition index (DI). First, 60 min insulinogenic index (IGI60) is calculated as (insulin60 min-insulin0 min[μU/mL])/(glucose60 min-glucose0 min [mmol/L]), using 0 min and 60 min values of OGTT. Then DI is calculated by multiplying IGI60 with composite ISI to reflect beta-cell function adjusting for the insulin sensitivity. DI will be evaluated at baseline and every 6 months until 12 months of GAHT.
Change from Baseline Bone Mineral Density at 12 months | 12 months
  Bone mineral densities (g/cm^2) of lumber spine and hip will be evaluated by dual-energy X-ray absorptiometry at baseline and 12 months of GAHT.
Depression Changes from Baseline Psychological Questionnaires at 12 months | 12 months
  Patient Health Questionnaire will be tested at baseline and every 3 months until 12 months to understand the effects of GAHT
Anxiety Changes from Baseline Psychological Questionnaires at 12 months | 12 months
  Generalized anxiety disorder scale will be tested at baseline and every 3 months until 12 months to understand the effects of GAHT
Suicide Ideation Changes from Baseline Psychological Questionnaires at 12 months | 12 months
  Beck scale for suicide ideation will be tested at baseline and every 3 months until 12 months to understand the effects of GAHT
Gender Dysphoria Changes from Baseline Psychological Questionnaires at 12 months | 12 months
  Utrecht gender dysphoria scale will be tested at baseline and every 3 months until 12 months to understand the effects of GAHT
Social Exclusion Changes from Baseline at 12 months | 12 months
  Cyberball task will be tested at baseline and every 3 months until 12 months to understand the effects of GAHT.
Functional brain Change after 6 months of GAHT | 6 months
  Change of functional connectivity will be analyzed to understand at 6 months of GAHT.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 12 months
  The incidence of adverse events during the 12 months of GAHT will be calculated, including thromboembolic events, drug-induced liver injury, hyperkalemia, newly diagnosed cardiovascular disease, erythrocytosis and newly diagnosed tumor.
Change from Baseline Body Mass Index at 12 months | 12 months
  Body mass index is calculated as [weight (kg) / height (m)^2], which will be evaluated at baseline and every 3 months until 12 months of GAHT.
Change from Baseline Waist-hip Ratio at 12 months | 12 months
  Waist-hip ratio is calculated as [waist (cm)/hip (cm)], which will be evaluated at baseline and every 3 months until 12 months of GAHT.
Change from Baseline Body Composition at 12 months | 12 months
  Fat percentage (%) and lean mass (kg) will be assessed using the InBody S10. The body composition will be evaluated at baseline and 12 months of GAHT.
Change from Baseline Breast Volume of transgender women at 12 months | 12 months
  Breasts of transgender women will be shot in 360° with 3D photography. The volume (ml) of both sides will be measured by the image analysis at baseline and every 6 months until 12 months of GAHT.
Change from Baseline Homeostatic Model Assessment Index (HOMA-IR) at 12 months | 12 months
  HOMA-IR is calculated as [(fasting insulin [µU/mL] × fasting glucose [mmol/L])/22.5]. HOMA-IR will be evaluated at baseline and every 6 months until 12 months of GAHT.
Change from Baseline Homeostatic Model Assessment of Beta-cell function (HOMA-β) at 12 months | 12 months
  HOMA-β is calculated as [20 × (fasting insulin [μU/mL]) × (fasting glucose -3·5 [mmol/L])]. HOMA-β will be evaluated at baseline and every 6 months until 12 months of GAHT.
Change from Baseline Serum Uric Acid at 12 months | 12 months
  Serum Uric Acid levels (μmol/l) will be evaluated at baseline and every 3 months until 12 months of GAHT.
Comparison of Transgender and Cisgender Functional Brain Patterns | At baseline
  Functional connectivity will be compared at baseline to understand the brain patterns of transgender.
Comparison of Transgender and Cisgender Cognitive Ability | At baseline
  Performance of mental rotation task of transgender and cisgender will be compared at baseline to understand the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Tianpei Hong, PhD., M.D., Principal Investigator — Department of Endocrinology and Metabolism, Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Dataset is available from the corresponding author on reasonable request.